CLINICAL TRIAL: NCT07221955
Title: The Impact of Qualia Gluthathione+ on Blood Glutathione Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qualia Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: QLS-019
Record Dates: First submitted 2025-10-24; First posted 2025-10-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Effects of Qualia Glutathione+ on Blood Glutathione Levels; Glutathione

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Qualia Glutathione+ version 1 (Active Comparator): Qualia Glutathione+ version 1 manufactured by Qualia Life Sciences
  Interventions: Dietary Supplement: Qualia Glutathione+ version 1
- Qualia Glutathione+ version 2 (Active Comparator): Qualia Glutathione+ version 2 manufactured by Qualia Life Sciences
  Interventions: Dietary Supplement: Qualia Glutathione+ version 2
- Placebo (Placebo Comparator): Rice flour placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Qualia Glutathione+ version 1 — Qualia Glutathione+ version 1 manufactured by Qualia Life Sciences
  Arms: Qualia Glutathione+ version 1
Dietary Supplement: Qualia Glutathione+ version 2 — Qualia Glutathione+ version 2 manufactured by Qualia Life Sciences
  Arms: Qualia Glutathione+ version 2
Dietary Supplement: Placebo — Rice flour
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group, triple-armed, study evaluating the effects of two distinct Qualia Glutathione+ formulations on Whole Blood Glutathione levels in the blood of healthy adults aged 45-75 years. Approximately 18 participants will be randomized to one of three study arms: Qualia Glutathione+ version 1, Qualia Glutathione+ version 2, or placebo. Each participant will take two or three capsules of their assigned product once daily in the morning, with or without food, over a 20-day period. The primary outcome is the change in blood glutathione levels, assessed via in lab blood collection at baseline and study completion. Secondary endpoints include questionnaires measuring health-related quality of life, fatigue, and cognitive functioning (PROMIS Global Health-10, PROMIS Short Form v1.0 - Fatigue 10a, PROMIS Cognitive Function - Short Form 8a), evaluation of safety and tolerability, and an Overall Experience Questionnaire (Appendices 1, 4-7). All assessments, including electronic questionnaires, are completed remotely without in-person visits.

ELIGIBILITY:
Inclusion criteria:

* Provide voluntary, written, informed consent to participate in the study
* Agree to provide a valid cell phone number and are willing to receive communications through text
* Can read and write English
* Willing to not begin taking any new supplements during the study and continue taking any supplements they are currently using regularly
* Willing to complete questionnaires, records, and diaries associated with the study.
* Healthy male and female participants aged 45-75 years
* Willing to go to a local blood draw location for a Whole Blood Total Glutathione measurement (baseline and Day 20)
* Willing to avoid starting new or stopping any existing dietary supplements throughout the study

Exclusion criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the trial
* Known food intolerances/allergy to any ingredients in the product
* Having any of the following conditions: Psychiatric conditions, neurologic disorders, endocrine disorders, cancer
* Having had a significant cardiovascular event in the past 6 months
* Taking MAO inhibitors, SSRIs, or any other psychiatric or neurological medicines
* On immunosuppressive therapy
* Adults lacking capacity to consent
* Active Smokers
* Diagnosed Diabetics

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-12-02 (Estimated); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Total Glutathione levels from baseline to Day 20 | 0-20 days
  To assess between-group differences in the change in blood Total Glutathione levels from baseline to Day 20 following supplementation with Qualia Glutathione version 1 versus placebo and Qualia Glutathione version 2 versus placebo

SECONDARY OUTCOMES:
between-group differences in blood Total Glutathione levels | baseline to day 20
  To assess the between-group differences in blood Total Glutathione levels from baseline to Day 20 following supplementation between Qualia Glutathione version 1 and Qualia Glutathione version 2.
within-group differences in the change in blood Glutathione levels | baseline to day 20
  To assess within-group differences in the change in blood Glutathione levels
Safety and Tolerability survey | baseline to days 7, 14 and 20
  To evaluate side effect profiles using a custom Safety and Tolerability survey.
PROMIS Global Health-10 | baseline to days 7, 14 and 20
  The PROMIS® Global Health Scale v1.2 (also known as the PROMIS-GH or PROMIS-10) is a 10-item, non-disease-specific questionnaire for adults to assess general physical and mental health. It yields two main scores, a Global Physical Health (GPH) T-score and a Global Mental Health (GMH) T-score, derived from four items each, to understand overall health perceptions. The scale is widely translated and free for use in clinical and research settings.
  * Raw Score Minimum and Maximum: 0-20
  * The higher the score, the better
PROMIS Short Form v1.0 - Fatigue 10a | baseline to days 7, 14 and 20
  The PROMIS Fatigue item banks assess a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. The fatigue short forms are universal rather than disease-specific. All assess fatigue over the past seven days.
  Raw Score Minimum and Maximum: 10-50 the lower the better
PROMIS Cognitive Function - Short Form 8a | baseline to days 7, 14 and 20
  The PROMIS Cognitive Function v2.0 - Short Form 8a is an 8-item self-report questionnaire designed to assess perceived cognitive function over the past seven days. It measures difficulties in areas such as forming thoughts, concentration, attention, thinking speed, memory, and the ability to shift between tasks.
  - Raw Score Minimum and Maximum: 8-40 - The higher the score, the better

CONTACTS AND LOCATIONS:
Locations (1):
- Qualia Life Sciences, Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: No